CLINICAL TRIAL: NCT06325098
Title: Implementation of a Diagnostic Workflow for Personalized Diagnosis of Nephrotic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Paola Romagnani, Professor, MD, PhD, Meyer Children's Hospital IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PER-NEPH
Record Dates: First submitted 2024-03-01; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Intervention Model Description: Patients with nephrotic syndrome (SSNS, SRNS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with SSNS (Experimental): Patients with SSNS and patients undergoing renal transplantation for NS with post-transplant disease recurrence will be enrolled for serum sampling for the study of immunological and/or permeabilizing factors (including anti-nephrin antibodies).
  Interventions: Diagnostic Test: Anti-nephrin antibodies
- Patients with SRNS undergoing genetic testing by WES (Experimental): Patients with SRNS undergoing genetic testing by WES and variant prioritization will undergo serum sampling for the study of immunologic and/or permeabilizing factors (including the anti-nephrin antibodies), and urine sampling for u-RPC cultures.
  Interventions: Diagnostic Test: Anti-nephrin antibodies; Diagnostic Test: u-RPC cultures

INTERVENTIONS:
Diagnostic Test: Anti-nephrin antibodies — Assessment of anti-nephrin antibodies on serum samples and in vitro study of permeabilizing effect on 3D organ-on-a-chip models and STED microscopy on healthy human kidneys.
Diagnostic Test: u-RPC cultures — Urine sample collection for u-RPC cultures
  Arms: Patients with SRNS undergoing genetic testing by WES

SUMMARY:
Nephrotic syndrome (NS) is a clinical picture common to several diseases resulting from damage to podocytes and glomerular filtration barrier. Currently, there is limited consensus regarding the diagnostic pathway and management of the specific etiology. Some patients show complete response to first-line steroid therapy (steroid-sensitive nephrotic syndrome, SSNS), especially in children and young adults. The prognosis of this group is generally favorable. In contrast, patients unresponsive to steroids (steroid-resistant NS, SRNS) frequently undergo immunosuppressive therapies, which are burdened with numerous side effects. Resistance to treatment is associated with a high likelihood of progression to chronic renal disease (CKD) and kidney failure (ESKD). Recent evidence suggests that immunological mechanisms (including permeabilizing factors) are involved in the pathogenesis of post-transplant NS recurrence and SSNS.

Providing patients with NS with a correct diagnosis is the cornerstone of personalized medicine, reducing morbidity and side effects of therapies, ensuring their appropriate prescription, and slowing or preventing progression to ESKD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NS (SSNS, SRNS, or NS relapsed after transplantation regardless of initial response to steroid therapy)
* Age below 40 years at disease onset
* Availability of clinical information
* Signed informed consent form

Exclusion Criteria:

* Age at onset above 40 years
* Kidney biopsy proving lesions other than FSGS and MCD

Ages: 1 Month to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Role of anti-nephrin antibodies in the pathogenesis of NS | From enrollment until the last patient visit (up to 12 months from enrollment)
  The presence of circulating permeabilizing factors, including anti-nephrin antibodies, will be evaluated in serum samples of patients with NS and/or kidney transplant recipients with NS recurrence. The results will be correlated with the clinical history of disease in order to understand the disease pathomechanisms and the risk of recurrence.

SECONDARY OUTCOMES:
Functional role of VUS in the pathogenesis of SRNS | From enrollment until the last patient last visit (up to 12 months from enrollment)
  The functional role of VUS identified by WES will be assessed by in vitro studies on u-RPCs and 3D organ-on-a-chip models.
  The results will be expressed as diagnostic rate, i.e., number of conclusive diagnosis allowed by functional studies of VUS/number of patients enrolled in the study.
Identification of potential predictive biomarkers of renal outcome. | From enrollment until the last patient visit (up to 12 months from enrollment)
  The identification of potential biomarkers of disease progression and kidney failure will be performed by gene expression by scRNA-seq of u-RPCs. The results will be correlated to clinical data.
Cost-effectiveness analysis | From enrollment of the last patient until the last visit (up to 12 months from enrollment)
  A modeled cost-effectiveness analysis (including direct and indirect medical costs) will be performed to compare the proposed diagnostic algorithm with the current standard-of-care.

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital IRCCS, Florence, Italy

IPD SHARING:
Plan to Share IPD: No